CLINICAL TRIAL: NCT00076154
Title: CSP #500A - National Registry of Veterans With Amyotrophic Lateral Sclerosis
Brief Title: National Registry of Veterans With Amyotrophic Lateral Sclerosis and DNA Bank
Acronym: ALS Registry
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: ALS Association (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 500A
Record Dates: First submitted 2004-01-14; First posted 2004-01-16 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: ALS
Keywords: ALS

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples or blood or mouthwash were collected in veterans' homes by nurses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
This study will identify living veterans with amyotrophic lateral sclerosis (ALS) through a national registry that is being developed. Diagnosis of ALS will be verified by study neurologists via medical record review. Registry participation includes a bi-annual telephone interview to collect functional status data.

DETAILED DESCRIPTION:
Primary Objective: To identify as completely as possible all veterans with ALS and to collect data which will be available for approved studies examining the cause(s) of ALS.

Secondary Objective: To provide a mechanism for the VA to inform veterans with ALS about clinical trials and other studies for which they may be eligible.

Primary Outcomes: Identification of all living veterans with ALS.

Intervention: N/A

Study Abstract: Amyotrophic lateral sclerosis (ALS) is an adult-onset, rapidly fatal neuromuscular disease of unknown etiology. ALS is a disease of high priority to the VA, particularly due to ongoing concerns about the health of veterans who served in the Gulf War. Efforts are needed to systematically identify and track veterans with ALS. Accordingly, the Department of Veterans Affairs (VA) is developing a national registry of veterans diagnosed with ALS.

Research Design: The registry will not be designed to test specific hypotheses but will focus on comprehensive identification of veterans with ALS who may be eligible for other studies.

Methodology: Eligible participants will include all living veterans with a physician diagnosis of ALS. Veterans with possible ALS will be identified through VA medical records, the Veterans Benefits Administration (VBA), and self-referral. Neurologists with expertise in ALS will review veterans' medical records to verify the diagnosis and determine eligibility. Upon enrollment, veterans will be asked to complete a brief telephone interview. Registry participants will also be contacted by telephone biannually to assess health and functional status. The VA may notify registry participants about clinical trials for which they may be eligible. A Scientific Review Committee will evaluate all studies that request use of registry data and/or access to Registry participants.

Results: N/A

Impacts: The registry will provide the VA with a valuable mechanism for involving veterans in clinical trials and other studies that may yield improved outcomes for ALS. In addition, data gathered as a part of the registry has the potential to benefit not only veterans, but also the larger community of individuals with ALS.

ELIGIBILITY:
Inclusion Criteria:

Living veteran with ALS verified via medical record review.

Exclusion Criteria:

Veteran whose medial records did not verify an ALS diagnosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Living veterans with an ALS diagnosis verified by medical records.
Sampling Method: Probability Sample
Enrollment: 2121 (Actual)
Dates: Start 2003-01; Primary Completion 2007-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Help studies using dates and DNA collected to determine possible genetic factor. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Z. Oddone, MD MHSc, Study Chair — VA Medical Center
Locations (1):
- Durham VA Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Schmidt S, Allen KD, Loiacono VT, Norman B, Stanwyck CL, Nord KM, Williams CD, Kasarskis EJ, Kamel F, McGuire V, Nelson LM, Oddone EZ. Genes and Environmental Exposures in Veterans with Amyotrophic Lateral Sclerosis: the GENEVA study. Rationale, study design and demographic characteristics. Neuroepidemiology. 2008;30(3):191-204. doi: 10.1159/000126911. Epub 2008 Apr 18. PMID 18421219
- [Result] Allen KD, Kasarskis EJ, Bedlack RS, Rozear MP, Morgenlander JC, Sabet A, Sams L, Lindquist JH, Harrelson ML, Coffman CJ, Oddone EZ. The National Registry of Veterans with amyotrophic lateral sclerosis. Neuroepidemiology. 2008;30(3):180-90. doi: 10.1159/000126910. Epub 2008 Apr 18. PMID 18421218
- [Result] Khishchenko N, Allen KD, Coffman CJ, Kasarskis EJ, Lindquist JH, Morgenlander JC, Norman BB, Oddone EZ, Rozear MP, Sabet A, Sams L, Bedlack RS. Time to diagnosis in the National Registry of Veterans with Amyotrophic Lateral Sclerosis. Amyotroph Lateral Scler. 2010;11(1-2):125-32. doi: 10.3109/17482960802572681. PMID 19153849
- [Result] Kasarkis EJ, Dominic K, Oddone EZ. The National Registry of Veterans with Amyotrophic Lateral Sclerosis: Department of Veterans Affairs Cooperative Studies Program (CSP) #500a. Amyotroph Lateral Scler Other Motor Neuron Disord. 2004 Sep;5 Suppl 1:129-32. doi: 10.1080/17434470410019915. PMID 15512895
- [Result] Pastula DM, Coffman CJ, Allen KD, Oddone EZ, Kasarskis EJ, Lindquist JH, Morgenlander JC, Norman BB, Rozear MP, Sams LA, Sabet A, Bedlack RS. Factors associated with survival in the National Registry of Veterans with ALS. Amyotroph Lateral Scler. 2009 Oct-Dec;10(5-6):332-8. doi: 10.3109/17482960802320545. PMID 19922120